CLINICAL TRIAL: NCT07357350
Title: Effectiveness of Pain Management Interventions in Patients With Abdominal and Pelvic Cancer in a Tertiary Care Hospital: A Prospective Observational Study
Brief Title: Effectiveness of Pain Management Interventions in Patients With Abdominal and Pelvic Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Ali Sarfraz Siddiqui, Associate Professor, Aga Khan University
Other Study IDs: 2025-12177-38695
Record Dates: First submitted 2026-01-15; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Abdominal Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective observational study is to observe the effectiveness of pain management interventions in patients with abdominal and pelvic cancer pain.

The main question[s] it aims to answer are:

* The effectiveness of pain management interventions.
* The frequency of pain intervention procedures and side effects and complications of pain management interventions

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic pain due to abdominal and pelvic cancer
* Both Male and Female
* Ages18-65 years
* Patients who with recurrence or metastasis

Exclusion Criteria:

* Patients who refuse to give consent
* Patients who were lost to follow up after initial visit or assessment
* History of severe depression or psychiatric illness
* History of surgical procedure due to cancer
* Patients with DNR code

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain due to abdominal and pelvic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-16 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient reported NRS score | First visit and then at 3 months
  Numeric Rating Score from 0 (no pain)- 10 (severe pain)

SECONDARY OUTCOMES:
Number of patients | From 2 weeks to 3 months.
  Number of patients on whom the intervention is performed.

IPD SHARING:
Plan to Share IPD: No